CLINICAL TRIAL: NCT00446394
Title: Exercise & Health Promotion for MCI: A Controlled Trial
Brief Title: Exercise and Activities for Independent Living With Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Linda Teri, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30692-J; 2R01AG014777 (NIH); IA0100 (Other: UW); 06-3067-C (Other: UW HSD old IRB application #)
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: cognition disorder; functional ability; psychomotor function; psychopathology; quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Cognition Disorders | interventions — Health Resources; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Resources and Activities for Life Long Independence (RALLI)
- 2 (Active Comparator)
  Interventions: Behavioral: Social Walking program (SW)

INTERVENTIONS:
Behavioral: Resources and Activities for Life Long Independence (RALLI) — Strengthening exercises, encouragement to walk daily, pedometer reading, health promotion information for 1.5 hours weekly for 9 weeks
  Arms: 1
Behavioral: Social Walking program (SW) — Group support for walking, pedometer reading, 1 hour weekly for 9 weeks
  Arms: 2

SUMMARY:
The purpose of this project is to evaluate an exercise and health promotion program for older adults with mild memory loss. The study will investigate the efficacy of a memory-enhanced exercise and health promotion program to determine whether it is more effective than a social walking program in delaying further memory decline, improving mood and physical function, and enhancing quality of life.

DETAILED DESCRIPTION:
This project is a randomized controlled trial to evaluate the efficacy of a group exercise and health promotion program designed specifically for older adults with Mild Cognitive Impairment (MCI). This study builds upon previous studies designed for cognitively intact older adults, with a supplemental study using a modified intervention for MCI participants, and for individuals with Alzheimer's disease.

Taken together, these prior investigations support the efficacy of behaviorally based exercise interventions in improving cognitive, physical, and affective status in cognitively intact and demented older adults. Results from a feasibility study suggest that these positive outcomes can also be obtained in older adults with MCI.

The current study will investigate the efficacy of the modified exercise program called RALLI (Resources and Activities for Life Long Independence) to determine whether it is more effective than the control condition, a social walking program (SW), in delaying cognitive decline, improving self-rated health and health behaviors, improving affect and physical function, and enhancing quality of life. The long-term efficacy of RALLI to delay conversion of MCI to dementia, reduce physical disability, maintain independent living, and improve physiological health indicators will also be investigated.

One hundred seventy participants over the age of 70 who meet American Academy of Neurology criteria for MCI will be recruited from independent living retirement residences. Participants will be randomly assigned to one of the two conditions (RALLI and SW) and assessed at baseline, post treatment (3 months), and follow up visits every 6 months for a total of 3 years (months 6, 12, 18, 24, 30, and 36). The hypothesis is that RALLI participants will experience better post-treatment outcomes than SW participants, and that gains will be maintained over 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment defined as
* - Memory complaint
* - Objective memory impairment for age and education
* - Largely intact general cognitive function
* - Essentially preserved activities of daily living
* - Not already diagnosed with dementia
* Insufficient physical activity defined as less than 150 minutes per week of moderate intensity physical activity
* Not currently in an exercise program similar to the study program

Exclusion Criteria:

* Not ambulatory
* Expected to move from the study geographic area during the study period
* Have a known terminal illness
* Actively suicidal, hallucinating, or delusional
* Hospitalized for a psychiatric disorder in the 12 months before baseline
* Uncontrolled chronic conditions, e.g. uncontrolled hypertension, unstable angina, uncontrolled blood glucose
* Blind or deaf

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive status | baseline, 3, 6, 12, 18, 24, 30, and 36 months

SECONDARY OUTCOMES:
Changes in health, affective, and functional status | baseline, 3, 6, 12, 18, 24, 30, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Teri, PhD, Principal Investigator — University of Washington School of Nursing
Locations (1):
- Northwest Research Group on Aging, Department of Psychosocial and Community Health, University of Washington School of Nursing, Seattle, Washington, United States